CLINICAL TRIAL: NCT05634512
Title: Evaluation of Intravenous Laronidase Pharmacokinetics Before and After Hematopoietic Cell Transplantation in Patients With Mucopolysaccharidosis Type IH.
Status: Active, not recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2021LS144; NCI-2022-09774 (Registry Identifier: NCI Trial ID); MT2021-29 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic Cell Transplantation; Mucopolysaccharidosis Type I
Keywords: MPS I; HCT
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Collect blood from patients with MPS-IH) undergoing laronidase therapy and stem cell transplant.: The primary aim is to characterize the PK of IV laronidase in individuals with MPS IH and identify patient specific covariates that impact drug exposure. The secondary aim is to identify key differences pre-and post-HCT leading to variability in PK parameters for patients receiving IV laronidase therapy for the treatment of MPS-IH.
  Interventions: Drug: Laronidase therapy and a stem cell transplant

INTERVENTIONS:
Drug: Laronidase therapy and a stem cell transplant — To identify key differences leading to variability in PK parameters for patients receiving IV laronidase therapy for the treatment of MPS-IH. There will be 12 samples per patient (6 pre-transplant and 6-post-transplant). Laronidase will be administered IV per protocol using standard dosing (0.58 mg/kg intravenously on a weekly basis), and six (n=6) blood samples will be collected over 24 hours for the determination of mononuclear cell lysates and plasma laronidase concentrations for a total of 18mL. The second PK monitoring will be obtained using the same PK design but following complete or near-completedonor derived myeloid engraftment which is evaluated at different time pointspost-HCT (day 30, day 42, day 60). The standard is to continue ERT through 8 weeks post-transplant.

SUMMARY:
This is a prospective, observational multicenter study to collect blood from patients with mucopolysaccharidosis type IH undergoing laronidase therapy and a stem cell transplant.

Sixteen patients will be enrolled over a 24 month period.

ELIGIBILITY:
Inclusion Criteria:

* Between 0 to 3 years of age

  * Meet protocol specific eligibility criteria for allogeneic HCT for MPS IH
  * Planning to receive laronidase both pre and post-transplant in an inpatient setting as part of standard-of-care treatment. Virtually all patients with MPSIH being considered for transplantation at the University of Minnesota are already receiving enzyme infusions, and it is standard practice to continue to give enzyme infusions to 8 weeks post-transplant. Therefore, participation will not modify the treatment course.

Exclusion Criteria:

* Patient's parent/ legal guardians are unable to provide informed consent.

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study entry is open to pediatric patients regardless of gender or ethnic background. While there will be every effort to seek out and include females and minority patients, the patient population is dependent upon the MPS-IH populations at the University of Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Identify covariates that impact drug exposure | 2 years
  Measure indicators for body size and maturation contribute to variability in laronidase exposure in patients with MPS IH.
Identify key differences pre- and post-HCT leading to variability in PK parameters | 2 years
  Measure endogenous source of enzyme present in relation to the transplanted cells.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, Principal Investigator — University of Minnesota Masonic Cancer Center
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No